CLINICAL TRIAL: NCT05309512
Title: A Phase Ia/Ib Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics/Pharmacodynamics, and Antitumor Activity of KN052 in Chinese Subjects With Advanced Solid Tumors
Brief Title: Clinical Study of KN052 in Chinese Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on the differentiated R&D strategy, the sponsor applies for the termination of the project.
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN052-CHN-001
Record Dates: First submitted 2022-03-09; First posted 2022-04-04 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2023-07

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KN052 single drug group (Experimental): The 8 dose groups in the dose increasing period were intravenous administration of 0.01mg/kg, 0.1mg/kg, 0.3mg/kg, 1mg/kg, 2mg/kg, 4mg/kg, 6mg/kg and 9mg/kg every two weeks, respectively. Based on the selected maximum tolerated dose of Q2W and in combination with the pharmacokinetic model, the sponsor would consider adding 1-2 Q3W treatment groups, with 6-12 patients in each dose group for DLT observation to explore the optimal dose regimen. The queue extension period is dose RP2D; Give it intravenously every two weeks or three weeks.
  Interventions: Biological: KN052

INTERVENTIONS:
Biological: KN052 — 0.01mg/kg, 0.1mg/kg, 0.3mg/kg, 1mg/kg, 2mg/kg, 4mg/kg, 6mg/kg, 9mg/kg, RP2D once every two or three weeks intravenously

SUMMARY:
This is a phase Ia/Ib open, multicenter study of solid tumor subjects in China.Including dose increasing period and cohort expansion period.A BOIN design is used in the dose escalation phase,a total of 8 dose groups were designed.In the expansion phase of the cohort, 15 to 30 subjects will be enrolled in a specific tumor type (liver cancer, stomach cancer, kidney cancer, melanoma, urothelial carcinoma, and other tumors determined by the SMC).

ELIGIBILITY:
Inclusion Criteria:

1. The subject can understand the informed consent, participate in and sign the informed consent voluntarily;
2. Subjects are at least 18 years old and <80 years old on the day of signing the informed consent, male or female, and are willing to follow the study procedures;
3. Solid tumors were confirmed histologically or cytologically. Subjects in the dose escalation phase were late unresectable or metastatic entities Patients with cancer must have received standard care and have no other standard care options with a proven survival benefit; or Subjects with refractory solid tumors who could not tolerate or had contraindications to standard treatments, including chemotherapy, Targeted therapy;
4. Measurable lesions at baseline according to RECIST 1.1; If subject has only 1 measurable disease at baseline The lesion area must not have received previous radiotherapy, or there is evidence of significant progression of the lesion after the end of radiotherapy;
5. ECOG score 0 or 1;
6. The laboratory test met the standard within 7 days before the first administration;
7. Life expectancy ≥3 months;
8. Fertile female subjects must have a negative serum pregnancy test within 7 days prior to first dosing;
9. Fertile female subjects or fertile male subjects with a partner agree to use highly effective contraception beginning 7 days before first dosing (annual failure rate less than 1%) until 24 weeks after completion of dosing.

Exclusion Criteria:

1. Subjects with untreated active BMS; Subjects with pia meningeal metastasis;
2. Received any other medication within 28 days prior to administration or 5 half-lives, whichever is shorter, but at least 2 weeks Interventional clinical trial therapy or other systemic chemotherapy, immunotherapy, targeted therapy and endocrine therapy;
3. Major surgery (transabdominal, transthoracic, etc.) was performed within 28 days prior to administration; Not including diagnosis Sexual puncture or peripheral vascular access replacement);
4. Had received radical radiotherapy within 3 months before administration in this study; 2 weeks prior to administration of palliative radiotherapy and radiotherapy are permitted Dose in line with local standards for palliative care;
5. Systemic corticosteroid (≥10 mg/ day prednisone, or other corticosteroid equivalent) or immunosuppressant treatment is required for 7 consecutive days within 14 days prior to the first administration of the drug in this study;
6. Received live vaccine (including live attenuated vaccine) within 28 days prior to administration;
7. Past or current interstitial pneumonia/lung disease requiring systematic hormone therapy;
8. Previous or current autoimmune diseases;
9. Other malignant tumors within 5 years prior to first administration;
10. Suffering from uncontrolled complications;
11. Toxicity of previous antitumor therapy did not return to CTCAE grade ≤1 (NCI-CTCAE V5.0) or baseline level;
12. Previous history of allogeneic bone marrow or organ transplantation;
13. In addition to anti-PD-(L)1 drugs or anti-CTLA-4 drugs, other antibodies/drugs (immune checkpoint) targeting T cell coregulatory proteins, such as OX40, 4-1BB,LAG3, TIM3, TIGIT or anti-CD127, have been used in the past;
14. Previous history of intolerance to anaphylaxis to antibody drugs (grade ≥3 NCI-CTCAE V5.0); Any speed before A history of allergic reactions or uncontrolled asthma; Significant prior drug allergy;
15. Pregnant and/or breastfeeding women;
16. Other conditions that may affect the safety or compliance of the drug treatment in this study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
MTD（ Maximum tolerated Dose） | Throughout the duration of the study，About 1 year
  MTD (Maximum tolerated Dose) is the dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate based on the BOIN Design
ORR（Objective Response Rate) | Throughout the duration of the study，About 1 year
  Objective response rate (ORR) was defined as the proportion of participants who achieve either complete response [CR] or partial response [PR] per Response Evaluation Criteria in Solid Tumors (RECIST v1.1）
DOR(Duration Of Response) | Throughout the duration of the study，About 1 year
  Defined as the time from the first evaluation of objective response to the first evaluation of PD or death from any cause prior to PD

SECONDARY OUTCOMES:
The probability of adverse events | Throughout the duration of the study，About 1 year
  Including the occurrence probability of TESAE, TEAE, TRAE, irAE, IRR and AE above grade CTCAE 3
Frequency of interruption, delay, and termination of dosing | Throughout the duration of the study，About 1 year
  The frequency of interrupted, delayed, and discontinued dosing was statistically analyzed by treatment dose group/cohort (tumor type)
Frequency of immunogenicity | Throughout the duration of the study，About 1 year
  Frequency of occurrence of anti-KN052 antibody and neutralizing antibody
Cmax of KN052 | Throughout the duration of the study，About 1 year
  Maximum observed serum concentration of KN052
Tmax of KN052 | Throughout the duration of the study，About 1 year
  Time of Maximum observed serum concentration (Tmax) of KN052
AUC(0-T) for KN052 | Throughout the duration of the study，About 1 year
  Adjusted geometric means of area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUC(0-T)) for KN052

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No